CLINICAL TRIAL: NCT03960424
Title: Diabetes Management Program for Hispanic/Latino
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-0002
Record Dates: First submitted 2019-05-09; First posted 2019-05-23 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes Mellitus; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Mixed Methods Design, incorporating adaptations before RCT trial commencement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Telemonitoring (DTM) (Experimental): Diabetes Telehealth Management (DTM), based on the 2018 ADA Standards for Type 2 Diabetes (T2D), uses smart devices to share information between patients, caregivers, and clinicians. DTM includes:1) weekly real time "virtual" visit between patient and clinician 2) vital signs monitoring/interpretation 3) diabetes management 4) patient interactive educational videos and "teach back" quizzes, reinforcing self-management strategies 5) a caregiver app with supportive capability.
  Interventions: Behavioral: Diabetes Telemonitoring
- Comprehensive Outpatient Management (COM) (Active Comparator): Comprehensive Outpatient Management (COM) is the most realistic evidence-based comparator, in that it is the most frequently recommended and used option for US T2D patients. COM, like DTM, is consistent with the 2018 American Diabetes Association (ADA) Standards which include, but are not limited to, past medical and family history, social history, medications, screening, physical examination, laboratory evaluation, etc.Patients are instructed to monitor blood glucose (within physician recommendations), and have routine or "well" visits every 3 months. Patients can set appointments with a T2D educator. COM patients will receive monthly calls from the study Registered Nurse (RN) to collect data.
  Interventions: Other: Comprehensive Outpatient Management

INTERVENTIONS:
Other: Comprehensive Outpatient Management — Patients receiving comprehensive outpatient management experience typical care received in the outpatient setting.
  Other Names: COM
  Arms: Comprehensive Outpatient Management (COM)
Behavioral: Diabetes Telemonitoring — Diabetes Telehealth Management (DTM), based on the 2018 ADA Standards for T2D, uses smart devices to share information between patients, caregivers, and clinicians.
  Other Names: DTM
  Arms: Diabetes Telemonitoring (DTM)

SUMMARY:
To compare Diabetes Telemonitoring to comprehensive outpatient management (COM) on critical patient-centered outcomes, including HbA1c.

DETAILED DESCRIPTION:
The investigators propose a multiphase mixed method, Comparative Effectiveness Research Randomized Control Trial (CER RCT) to:

Specific Aim 1: Assess usability of an evidence-based DTM intervention utilizing a Community Based Participatory Research (CBPR) approach and adapt it to facilitate acceptability and feasibility in a population of H/L patients with T2D, and their caregivers and providers.

Specific Aim 2: Assess whether H/L patients receiving DTM attain significantly improved patient-centered outcomes compared to COM, through a CER RCT. Expected outcomes include improved diabetes quality of life (QoL), glucose management (GM), blood pressure (BP), cholesterol, medication adherence, and diabetes self-efficacy (SE), and reduced diabetes distress, problem areas in diabetes (PAID), inpatient utilization, unscheduled T2D physician visits and sick days.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic patients with a diagnosis of diabetes
* Speaks English or Spanish

Exclusion Criteria:

* Patient is not Hispanic
* Patient does not have a diagnosis of diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | 6 months
  HbA1c

SECONDARY OUTCOMES:
HbA1c | 12 months
  Hemoglobin A1c
Hypoglycemia episodes | 6 months
  Number of hypoglycemia episodes
Adherence | 6 months
  Adherence to Refills and Medications - Diabetes (ARMS-D)
Diabetes self-efficacy | 6 months
  Diabetes Self-Efficacy Scale
PAID | 6 months
  Problem Areas in Diabetes Scale
Weight | 6 months
  lbs
Cholesterol | 6 months
  Changes in cholesterol over time
Blood Pressure | 6 months
  BP
Diabetes Quality of life | 6 months
  Diabetes-39 is a validated instrument specifically designed to measure quality of life for diabetes patients

CONTACTS AND LOCATIONS:
Overall Officials: Renee Pekmezaris, PhD, Principal Investigator — Feinstein Institute for Medical Research
Locations (1):
- Feinstein Institute of Medical Research, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pekmezaris R, Williams MS, Pascarelli B, Finuf KD, Harris YT, Myers AK, Taylor T, Kline M, Patel VH, Murray LM, McFarlane SI, Pappas K, Lesser ML, Makaryus AN, Martinez S, Kozikowski A, Polo J, Guzman J, Zeltser R, Marino J, Pena M, DiClemente RJ, Granville D. Adapting a home telemonitoring intervention for underserved Hispanic/Latino patients with type 2 diabetes: an acceptability and feasibility study. BMC Med Inform Decis Mak. 2020 Dec 7;20(1):324. doi: 10.1186/s12911-020-01346-0. PMID 33287815

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT03960424/Prot_SAP_004.pdf
  • Informed Consent Form (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT03960424/ICF_005.pdf